CLINICAL TRIAL: NCT01506167
Title: An Observational Study of Avastin® (Bevacizumab) in Combination With Chemotherapy for Treatment of First-line Metastatic Colorectal Adenocarcinoma
Brief Title: An Observational Study of Avastin (Bevacizumab) in Patients With Metastatic Colorectal Cancer (ACORN)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27971
Record Dates: First submitted 2012-01-05; First posted 2012-01-09 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; XELOX; Fluorouracil; Capecitabine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

GROUPS / COHORTS (7):
- Bevacizumab and Capecitabine/Oxaliplatin: Participants who receive bevacizumab in combination with capecitabine/oxaliplatin
  Interventions: Drug: Bevacizumab; Drug: Capecitabine/Oxaliplatin
- Bevacizumab and Fluorouracil/Folinic Acid/Oxaliplatin: Participants who receive bevacizumab in combination with fluorouracil/folinic acid/oxaliplatin
  Interventions: Drug: Bevacizumab; Drug: Fluorouracil/Folinic Acid/Oxaliplatin
- Bevacizumab and Capecitabine: Participants who receive bevacizumab in combination with capecitabine
  Interventions: Drug: Bevacizumab; Drug: Capecitabine
- Bevacizumab and Fluorouracil/Folinic Acid/Irinotecan: Participants who receive bevacizumab in combination with fluorouracil/folinic acid/irinotecan
  Interventions: Drug: Bevacizumab; Drug: Fluorouracil/Folinic Acid/Irinotecan
- Bevacizumab and Capecitabine/Irinotecan: Participants who receive bevacizumab in combination with capecitabine/irinotecan
  Interventions: Drug: Bevacizumab
- Bevacizumab and Fluorouracil +/- Folinic Acid: Participants who receive bevacizumab in combination with fluorouracil +/- folinic acid
  Interventions: Drug: Bevacizumab; Drug: Fluorouracil +/- Folinic Acid
- Other: Participants who receive bevacizumab in combination with other first-line chemotherapy regimens
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab was administered as part of standard first-line treatment
  Other Names: Avastin®
Drug: Capecitabine/Oxaliplatin — Capecitabine/oxaliplatin were administered along with bevacizumab as part of standard first-line treatment
  Groups: Bevacizumab and Capecitabine/Oxaliplatin
Drug: Fluorouracil/Folinic Acid/Oxaliplatin — Fluorouracil/folinic acid/oxaliplatin were administered along with bevacizumab as part of standard first-line treatment
  Groups: Bevacizumab and Fluorouracil/Folinic Acid/Oxaliplatin
Drug: Capecitabine — Capecitabine was administered along with bevacizumab as part of standard first-line treatment
  Groups: Bevacizumab and Capecitabine
Drug: Fluorouracil/Folinic Acid/Irinotecan — Fluorouracil/folinic acid/irinotecan were administered along with bevacizumab as part of standard first-line treatment
  Groups: Bevacizumab and Fluorouracil/Folinic Acid/Irinotecan
Drug: Fluorouracil +/- Folinic Acid — Fluorouracil +/- folinic acid were administered along with bevacizumab as part of standard first-line treatment
  Groups: Bevacizumab and Fluorouracil +/- Folinic Acid

SUMMARY:
This prospective, multi-center, observational study will assess the safety and efficacy of Avastin (bevacizumab) in daily practice in patients with metastatic colorectal cancer who have received no previous treatment for advanced disease and are receiving Avastin in combination with a standard of care first-line chemotherapy regimen. Data will be collected for 1.5 years or until death.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal cancer with no previous systemic treatment for advanced disease
* Receiving Avastin in combination with a first-line standard of care chemotherapy regimen
* Avastin initiated at the same time as first-line chemotherapy regimen

Exclusion Criteria:

* Investigational, non-standard of care first-line chemotherapy regimen for treatment of metastatic colorectal cancer
* Contraindication to Avastin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with metastatic colorectal cancer
Sampling Method: Probability Sample
Enrollment: 719 (Actual)
Dates: Start 2012-07-06 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2017-03-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Serious Adverse Events (SAEs) | 1.5 years
  An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires new in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is a significant medical event in the investigator's judgment or requires intervention to prevent one or other of these outcomes.
Percentage of Participants with Grade 3-5 Avastin Related Adverse Events | 1.5 years
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, regardless of causal attribution. Adverse events were graded according to NCI-CTCAE, v4.0 (National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0).
Progression-Free Survival | 1.5 years
  Progression-Free Survival (PFS) was defined as the number of days from start of first-line therapy administration (earliest date of either the start of chemotherapy regimen administration or the start of Avastin) to the date of first occurrence of investigator-assessed disease progression or death. PFS was assessed using Kaplan-Meier method.
Overall Survival | 1.5 years
  Overall Survival (OS) is defined as the number of days from the start of first-line therapy (earliest date of either the start of chemotherapy regimen administration or the start of Avastin) to death by any cause.

SECONDARY OUTCOMES:
Percentage of Participants with Avastin Related Adverse Events of Special Interest | 1.5 years
  Adverse events of special interest (AESIs) are defined by their possible association with Avastin® treatment. The adverse events of special interest in this study include all grades of gastrointestinal perforation, fistulae, arterial and venous thromboembolic events, congestive heart failure and pulmonary haemorrhages; and Grade 2-5: hypertension, wound healing complications, proteinuria and mucocutaneous haemorrhages.
Reasons for Discontinuation of Avastin | 1.5 years
Median Progression Free Survival from Four Avastin Studies | 1.5 years (ACORN)
  PFS was defined as the number of days from start of first-line therapy administration (earliest date of either the start of chemotherapy regimen administration or the start of Avastin) to the date of first occurrence of investigator-assessed disease progression or death. The BRITE, BEAT and ARIES trials were conducted outside of the UK unlike the ACORN trial which was conducted in England only. Median PFS is presented for data from other registration trials and similar observational studies.
Median Overall Survival from Four Avastin Studies | 1.5 years (ACORN)
  OS is defined as the number of days from the start of first-line therapy (earliest date of either the start of chemotherapy regimen administration or the start of Avastin) to death by any cause. The BRITE, BEAT and ARIES trials were conducted outside of the UK unlike the ACORN trial which was conducted in England only. Median OS is presented for data from other registration trials and similar observational studies.
Percentage of Participants with Comparative AEs from Four Avastin® Studies | 1.5 years (ACORN)
  Comparative AEs included Gastrointestinal perforation; Haemorrhage (specific grade); All Haemorrhages; Hypertension; and Arterial thromboembolic events (cerebrovascular accident, myocardial infarction, transient ischaemic attack and other). The specific grade of haemorrhage was 3/4 for BRITE, 3/4 for BEAT and 3-5 for ARIES. The specific grade for ACORN was unknown. The BRITE, BEAT and ARIES trials were conducted outside of the UK unlike the ACORN trial which was conducted in England only.
Median Age of Participants in Four Avastin® Studies | Baseline
  The BRITE, BEAT and ARIES trials were conducted outside of the UK unlike the ACORN trial which was conducted in England only.
Percentage of Participants Over (or equal to) 75 Years of Age in Four Avastin Studies | Baseline
  The BRITE, BEAT and ARIES trials were conducted outside of the UK unlike the ACORN trial which was conducted in England only.
Percentage of Males and Females in Four Avastin Studies | Baseline
  The BRITE, BEAT and ARIES trials were conducted outside of the UK unlike the ACORN trial which was conducted in England only.
Eastern Cooperative Oncology Group (ECOG) Performance Status in Four Avastin Studies | 1.5 years (ACORN)
  ECOG Performance Status measured on-therapy (time between first dose and last dose date) assessed participant's performance status on 5 point scale: 0 is equal to (=) fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2=ambulatory (greater than [>] 50% of waking hours [hrs]), capable of all self care, unable to carry out any work activities; 3=capable of only limited self care, confined to bed/chair >50% of waking hrs; 4=completely disabled, cannot carry on any self care, totally confined to bed/chair; 5=dead. The BRITE, BEAT and ARIES trials were conducted outside of the UK unlike the ACORN trial which was conducted in England only.
Race/Ethnicity of Participants in Four Avastin Studies | Baseline
  The BRITE, BEAT and ARIES trials were conducted outside of the UK unlike the ACORN trial which was conducted in England only.
Percentage of Participants at Stage IV (at diagnosis) in Four Avastin Studies | Baseline
  The BRITE, BEAT and ARIES trials were conducted outside of the UK unlike the ACORN trial which was conducted in England only.
Percentage of Participants that Received Previous Systematic Treatment for CRC in Four Avastin Studies | Baseline
  The BRITE, BEAT and ARIES trials were conducted outside of the UK unlike the ACORN trial which was conducted in England only.
Sites of CRC in Four Avastin Studies | Baseline
  The BRITE, BEAT and ARIES trials were conducted outside of the UK unlike the ACORN trial which was conducted in England only.
Percentage of Participants with Primary Resection in Four Avastin Studies | Baseline
  The BRITE, BEAT and ARIES trials were conducted outside of the UK unlike the ACORN trial which was conducted in England only.
Metastatic Sites of CRC in Four Avastin Studies | Baseline
  The BRITE, BEAT and ARIES trials were conducted outside of the UK unlike the ACORN trial which was conducted in England only.
Ongoing Patient Medical Conditions in Four Avastin Studies | Baseline
  The BRITE, BEAT and ARIES trials were conducted outside of the UK unlike the ACORN trial which was conducted in England only.
Weeks of Further Treatment After 1st Line Chemotherapy | From disease progression until end of study.
  Number of weeks of further chemotherapy regimen administered after 1st line treatment.
Quality of Life as Assessed by the Euro-Quality of Life-5 Dimensions (EQ-5D) Weighted Index Score | Baseline and 3, 6, 9, 12, 15, 18, 21, 24 and 27 Months post chemotherapy
  The EQ-5D is composed of 5 single-item measures where participants responded to questions assessing health status by responding with either "no problems", "slight problems", "moderate problems", "severe problems" or "extreme [problem]/unable to perform" in the following categories: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Based on population surveys, an algorithm was used to combine the responses to each of these 5 measures into 1 single EQ-5D weighted index score ranging from -0.59 (extreme problems) to +1 (no problems) where a negative value indicated a worsening of perceived quality of life and a positive value indicated an improvement of perceived quality of life.
Quality of Life as Assessed by the Euro-Quality of Life-5 Dimensions (EQ-5D) Crosswalk Index Score | Baseline and 3, 6, 9, 12, 15, 18, 21, 24 and 27 Months post chemotherapy
  The EQ-5D is composed of 5 single-item measures where participants responded to questions assessing health status by responding with either "no problems", "slight problems", "moderate problems", "severe problems" or "extreme [problem]/unable to perform" in the following categories: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Based on population surveys, an algorithm was used to combine the responses to each of these 5 measures into 1 single EQ-5D index score ranging from -0.59 (extreme problems) to +1 (no problems) where a negative value indicated a worsening of perceived quality of life and a positive value indicated an improvement of perceived quality of life.
Response to the Burden of Illness Question: In the last three months how many times have health care professionals been to your home? | Baseline and 3, 6, 9, 12, 15, 18, 21, 24 and 27 Months post chemotherapy
Response to the Burden of Illness Question: In the last three months how many times have you seen health care professionals at your GP Surgery or day centre? | Baseline and 3, 6, 9, 12, 15, 18, 21, 24 and 27 Months post chemotherapy
Response to the Burden of Illness Question: In the last three months how many nights in total did you spend in hospital/hospice? | Baseline and 3, 6, 9, 12, 15, 18, 21, 24 and 27 Months post chemotherapy
Response to the Burden of Illness Question: In the last three months how many times did you visit the imaging department for these examinations? | Baseline and 3, 6, 9, 12, 15, 18, 21, 24 and 27 Months post chemotherapy
Response to the Burden of Illness Question: What was your employment status before diagnosis? | Baseline
Response to the Burden of Illness Question: What is your employment status now? | Baseline and 3, 6, 9, 12, 15, 18, 21, 24 and 27 Months post chemotherapy
Response to the Burden of Illness Question: Has your cancer resulted in you seeking support services? | Baseline and 3, 6, 9, 12, 15, 18, 21, 24 and 27 Months post chemotherapy
Response to the Burden of Illness Question: Has a previously employed family member had to take time off work to care for you? | Baseline and 3, 6, 9, 12, 15, 18, 21, 24 and 27 Months post chemotherapy
Response to the Burden of Illness Question: Has your cancer resulted in a family member seeking support? | Baseline and 3, 6, 9, 12, 15, 18, 21, 24 and 27 Months post chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (43):
- United Kingdom (43):
  - Royal United Hospital Bath; Diabetes and Lipid Research, Wolfson Centre, Bath
  - Wexham Park Hospital; Oncology, Berkshire
  - Queen Elizabeth Hospital, Birmingham
  - Birmingham Heartlands Hospital; Dept of Oncology, Birmingham
  - Bishop Auckland Hospital;Oncology Department, Bishop Auckland
  - University Hospital of North Staffordhire, Blackpool
  - Bradford Royal Infirmary; Dept of Medical Oncology C/O Ward15, Bradford
  - Bristol Haematology and Oncology Centre, Bristol
  - West Suffolk Hospital Nhs Trust; Gi Corridor, Bury St Edmunds
  - Kent & Canterbury Hospital, Canterbury
  - Cumberland Infirmary; Oncology Department, Carlisle
  - Broomfield Hospital; Oncology, Chelsmford
  - University Hospital North Tees, Cleveland
  - Castle Hill Hospital; Academic Oncology, Cottingham
  - Darlington Memorial Hospital, Darlington
  - Russells Hall Hospital; Dept of Hematology, Dudley
  - University Hospital of North Durham; Oncology, Durham
  - Harrogate Hospital, Harrogate
  - Northhwick Park Hospital;Oncology Department, Harrow
  - Ipswich Hospital; Oncology Pharmacy, Ipswich
  - Kidderminster Hospital; Oncology Dept, Kidderminster
  - Royal Free Hospital; Dept of Oncology, London
  - Guys Hosp./Med. Onc./3rd Fl. T; Clinical Trial Office, London
  - Queen Elizabeth Hospital, London
  - Macclesfield District General Hospital, Macclesfield
  - Maidstone & Tonbridge Wells Hospital; Kent Oncology Center, Maidstone
  - The James Cook University Hospital, Middlesbrough
  - Freeman Hospital, Newcastle upon Tyne
  - North Tyneside General Hospital, North Shields
  - Mount Vernon Cancer Centre, Northwood
  - Nottingham University Hospitals City Campus, Nottingham
  - Peterborough City Hospital, Edith Cavell Campus; Oncology Department, Peterborough
  - Derriford Hospital; Gastroenterology, Plymouth
  - Queen's Hospital, Romford
  - Scunthorpe General Hospital; Dept of Oncology, Scunthorpe
  - Stafford Hospital; Oncology Department, Stafford
  - The Royal Marsden Hospital, Sutton
  - Great Western Hospital, Swindon Cancer Research Unit; Osprey Unit Level 3, Swindon
  - Torbay Hospital; Oncology, Torquay
  - Royal Cornwall Hospital; Dept of Clinical Oncology, Truro
  - Walsall Manor Hospital, Walsall
  - Royal Hampshire County Hospital; Winchester & Andover Breast Unit, Winchester
  - The Royal Wolverhampton Hospitals NHS Trust, Wolverhampton

REFERENCES:
- [Derived] Khakoo S, Chau I, Pedley I, Ellis R, Steward W, Harrison M, Baijal S, Tahir S, Ross P, Raouf S, Ograbek A, Cunningham D; ACORN investigators. ACORN: Observational Study of Bevacizumab in Combination With First-Line Chemotherapy for Treatment of Metastatic Colorectal Cancer in the UK. Clin Colorectal Cancer. 2019 Dec;18(4):280-291.e5. doi: 10.1016/j.clcc.2019.07.003. Epub 2019 Jul 11. PMID 31451367